CLINICAL TRIAL: NCT07041255
Title: The First Prospective Randomized Trial Comparing Cold and Hot Loop Resection for Removal of Medium-sized Benign Colon Tumors in Moscow, Russia.
Brief Title: Comparison of Cold and Hot Loop Resection Techniques for the Removal of Medium-sized Benign Colon Tumors
Acronym: chs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06111985_02
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-01

CONDITIONS: Benign Colon Tumors
Keywords: cold snare resection; hot snare resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold EMR (Experimental): The time of removal, the number of fragments, complications, its immediate and remote results are assessed,histology result
  Interventions: Procedure: Cold endoscopic mucosal resection; Procedure: Hot endoscopic mucosal resection
- Hot EMR (Experimental): The time of removal, the number of fragments,
  , complications, and immediate and long-term results are assessed,histology result
  Interventions: Procedure: Cold endoscopic mucosal resection; Procedure: Hot endoscopic mucosal resection

INTERVENTIONS:
Procedure: Cold endoscopic mucosal resection — 3-4 ml of solution is injected into the submucosal layer under the formation. The formation with the surrounding mucous membrane (at least 1 mm from the edge of the formation) is captured with a specialized or standard polypectomy loop available to the operator (depending on the randomization result). The formation is removed by mechanical cutting without using electric current.
  Other Names: Cold EMR
Procedure: Hot endoscopic mucosal resection — 3-4 ml of solution is injected into the submucosal layer under the formation. The formation with the surrounding mucous membrane (at least 1 mm from the edge of the formation) is captured with a specialized or standard diathermic polypectomy loop available to the operator (depending on the randomization result). The formation is removed using electric current in the Endocat mode (or its analogue, providing alternating cutting and coagulation under the control of a processor built into the electrical unit).
  After the formation is removed, the resection site is examined in white light, then virtual chromoscopy (NBI), and then an examination with magnification. The examination results are recorded in the scientific protocol separately, and are assessed as a whole. The criteria for visual removal of the formation within healthy tissues are the absence of visible fragments of the formation. The time of complete cessation of capillary bleeding is recorded.
  Other Names: Hot EMR

SUMMARY:
Widespread introduction of high-resolution videocolonoscopy into clinical practice has led to an increase in the detection of epithelial lesions of the colon, a significant portion of which are small (<10 mm) and miniature (≤5 mm) lesions. According to the literature, 15.6-27% of colon lesions 6-9 mm in size and 4.4-10% of those ≤5 mm are high-risk lesions, i.e. they contain villous structures, foci of severe dysplasia or cancer. One of the methods for removing such lesions is the technique of cold loop polypectomy (CLP), i.e. mechanical removal of the polyp with a loop without the use of electric current. This method is common for colon lesions 4-9 mm in size. (For smaller lesions, a technically simple and effective method of removing them using biopsy forceps is most often used) Jung YS, Park JH, Kim HJ et al. Complete biopsy resection of diminutive polyps. Endoscopy 2013; 45: 1024-9). A number of studies have demonstrated the advantages of the CP technique over standard removal methods. "Cold" polypectomy reduces the incidence of complications associated with thermal effects on the mucous membrane and underlying tissues (Bo-In Lee. Polypectomy of Small Polyps: Technical Updates. IDEN 2016, 280-281). Not only the number of perforations and manifestations of postcoagulation syndrome is reduced (D. von Renteln1, H. Pohl. Polyp Resection - Controversial Practices and Unanswered Questions. Clin Transl Gastroenterol. 2017 Mar; 8(3): e76. doi: 10.1038/ctg.2017.6), but also delayed bleeding: 0% with cold snare removal versus 0.5-14% after classical removal using electric current (Horiuchi A, Nakayama Y et al. Removal of small colorectal polyps in anticoagulated patients: a prospective randomized comparison of cold snare and conventional polypectomy. Gastrointest Endosc. 2014 Mar;79(3):417-23. doi: 10.1016/j.gie.2013.08.040; T. Kawamura1, Y.Takeuchi A comparison of the resection rate for cold and hot snare polypectomy for 4-9 mm colorectal polyps: a multicentre randomised controlled trial (CRESCENT study) Gut Online First, published on September 28, 2017 as 10.1136/gutjnl-2017-314215) ! It is also important that the removal of polyps with a cold snare takes less time than with a hot one, averaging 18 min. versus 25 min. (Ichise Y1, Horiuchi A, Nakayama Y, Tanaka N. Prospective randomized comparison of cold snare polypectomy and conventional polypectomy for small colorectal polyps. Digestion. 2011;84(1):78-81. doi: 10.1159/000323959. However, there are currently clearly not enough large multicenter prospective randomized studies devoted to the comparison of the efficacy and safety of "standard" and cold polypectomy.

The opinion of specialists is also ambiguous regarding the instrumentation that should be used for endoscopic removal of small formations. Some endoscopists believe that the type of polypectomy snare used does not affect the efficacy, completeness and safety of removal of small formations, while others, on the contrary, pay special attention to the use of specially designed small-diameter snare loops, believing that only they are capable of ensuring the removal of formations in a single block in the vast majority of cases. (Horiuchi A, Hosoi K, Kajiyama M, et al. Prospective, randomized comparison of 2 methods of cold snare polypectomy for small colorectalpolyps. Gastrointest Endosc 2015;82:686-92.) The question of the need to inject fluid into the submucosal layer under the removed formation also requires a reasoned answer, given that many researchers skip this stage of the intervention and / or consider it unnecessary Toshiki Yamamoto, Sho Suzuki, Chika Kusano, Kyoko Yakabe, Maho Iwamoto, Hisatomo Ikehara, Takuji Gotoda, Mitsuhiko Moriyama. Histological outcomes between hot and cold snare polypectomy for small colorectal polyps. Saudi J Gastroenterol. 2017 Jul-Aug; 23(4): 246-252. doi: 10.4103/sjg.SJG_598_16

DETAILED DESCRIPTION:
Objective of the study: to prospectively compare the immediate, short-term and long-term results of cold and hot resection of the mucosa through a colonoscope, performed for non-invasive medium-sized (10-14 mm) epithelial lesions of the colon with a broad base.

Study objectives:

1. To evaluate the accuracy of high-resolution colonoscopy in white and narrow spectrum light with magnification in predicting the histological structure of medium-sized epithelial lesions of the colon with a broad base.
2. To conduct a comparative assessment of the completeness (in one block/in parts; R0/R1) and depth of resection of medium-sized epithelial lesions of the colon with a broad base according to endoscopic and morphological criteria.
3. To determine the comparative frequency of intra- and postoperative complications (bleeding, perforation, postcoagulation syndrome) during removal of medium-sized epithelial lesions of the colon with a broad base.

General characteristics of the clinical study. Design: prospective, randomized, controlled, single-center study.

It is planned to include at least 200 patients in the study until statistically significant indicators are obtained for all analyzed parameters, who will undergo Cold EMR or Hot EMR for one or more medium-sized (10-14 mm) non-invasive epithelial formations of the colon on a broad base.

Criteria for inclusion of patients:

1. Patient with one benign non-invasive epithelial formation of the colon of type Is and II, 10-14 mm in size
2. Age ≥ 18 years.
3. Signed informed voluntary consent for colonoscopy and removal of formations using the methods under study.

Exclusion criteria:

1. Reasonable suspicion of severe dysplasia/cancer, including with submucosal invasion based on the results of preoperative assessment (NICE - 3; JNET - 2b and 3; Kudo - Vi and Vn).
2. Colon formations less than 10 mm
3. Recurrent nature of the formation.
4. Presence of widespread malignant tumor in any part of the colon.
5. Use of other methods of endoscopic removal of the formation.
6. IBD.
7. Patient on hemodialysis
8. Uncorrectable coagulopathy (INR> 1.5).
9. Refusal to participate in the study.
10. General contraindications to endoscopic examination.

All patients will be randomly divided into 2 main groups using block stratification randomization: the Cold EMR Group and the Hot EMR Group. In addition, within each main group, the type of polypectomy loop will be randomly selected.

It is planned to evaluate the following patient characteristics:

1. Gender.
2. Age.
3. Taking aspirin (or analogues) and/or indirect anticoagulants
4. The degree of concomitant pathology, expressed in the concept of surgical-anesthesiological risk according to the ASA scale.
5. History of abdominal surgery
6. History of inflammatory diseases of the abdominal organs, including diverticulitis, usually leading to the formation of adhesions involving the colon,

The following study characteristics are planned to be assessed:

1. Nature of preparation (compliance/non-compliance with the recommended diet; drug(s) used, split preparation or not, time from the last dose to the start of colonoscopy), quality of preparation (according to the Boston scale).
2. Type of device used (HD? NBI? Possibility of magnification?)
3. Presence of sedation (Yes/No).
4. Use of a distal cap (Yes/No).
5. Use of an electromechanical pump

The following endoscopic characteristics of the epithelial lesion are planned to be assessed:

1. Localization (according to anatomical landmarks), preferably indicating the number of haustra from significant landmarks;
2. Size of the lesion (mm);
3. Type according to the Paris Classification of Epithelial Neoplasia;
4. Assessment of the surface microstructure according to NICE, JNET, WASP, Kudo.

The following characteristics of EMR are planned to be assessed:

1. Method of removal (Cold with injection of a solution into the submucosal layer or HLP with injection of a solution into the submucosal layer);
2. Type of current used in Hot EMR(Endocat).
3. Removal time (from the moment the loop is brought into the field of view until complete removal of the formation);
4. Method of removal (in fragments or as a single block);
5. Single loop closure (until complete cutting) or multiple (with tissue resistance)
6. Completeness of removal according to high-resolution endoscopy, virtual chromoscopy and magnification upon completion of the intervention (within healthy tissue/no)
7. Removal of the specimen (removed/lost) and the reason for loss
8. Use of prophylactic clipping (Yes/No) and indications for its use: deep post-resection defect (up to and including the muscle layer); perforation I have bowels; inability to achieve hemostasis; for social reasons (doctor, relatives, etc.)
9. Type and nature of adverse events (inability to cut the formation with a cold loop and the need for traction of a completely tightened loop to remove it; bleeding, perforation).

It is planned to evaluate the following characteristics in the postoperative period:

1. Presence of abdominal pain syndrome (Yes/No)
2. Temperature Yes/No (within 24 hours, above 37.2).
3. Type, time of occurrence, and nature of adverse events (bleeding, perforation, postcoagulation syndrome).
4. Type of observation after removal (outpatient/inpatient). If inpatient, for how long.
5. Compliance with a diet in the postoperative period (yes/no).
6. Use of antibiotics (yes/no).
7. Use of hemostatics (yes/no).

It is planned to evaluate the following morphological characteristics of the formation:

1. Fragmentation of the formation (yes/no)
2. Histological structure of the formation (examination of the removed specimen, according to the WHO and Vienna classification).
3. Quality of visualization of the resection boundaries in Cold EMR and Hot EMR (visualization: complete; difficult; impossible).
4. Morphological assessment of the completeness of removal (assessment of the specimen) - R0 - no cells of the formation along the resection line, R1 - there are cells of the formation along the resection line, Rx - the formation is removed in fragments or the status of the resection boundaries cannot be determined.
5. Presence of the muscularis mucosa in the sample (in % of the sample area).
6. Morphological assessment of the thickness of the submucosal layer and the diameter of the largest vessel in the specimen.

Technique of endoscopic intervention. To prepare for colonoscopy, it is recommended: to adhere to a low-residue diet for 2 days (the 3rd and 2nd days before the endoscopic intervention); the day before, drink only clear liquids; use full-volume PEG-based preparations (Fortrans) or a low-volume sulfate-based preparation (Eziclen) in split mode.

After visualizing the formation, its localization is assessed, its type according to the Paris classification of epithelial neoplasia, its size compared to the diameter of the catheter ("shirt") of the loop and the polypectomy loop itself in the open state. (If technically possible, the use of an endoscopic ruler is welcomed). The nature of the surface of the formation is assessed in white light and using virtual chromoscopy according to NICE, WASP; with magnification - according to JNET and, if necessary, according to Kudo with a 0.5-1.0% indigo carmine solution. If the selection criteria are met, randomization is performed and the formation is removed either by the CLP or HLP method.

Cold EMR technique. 3-4 ml of solution is injected into the submucosal layer under the formation. The formation with the surrounding mucous membrane (at least 1 mm from the edge of the formation) is captured by a specialized or standard polypectomy loop available to the operator (depending on the randomization result). The formation is removed by mechanical cutting without using electric current.

Hot EMR technique. 3-4 ml of solution is injected into the submucosal layer under the formation. The formation with the surrounding mucous membrane (at least 1 mm from the edge of the formation) is captured by a specialized or standard diathermic polypectomy loop available to the operator (depending on the randomization result). The formation is removed using electric current in the Endocat mode (or its analogue, providing alternating cutting and coagulation under the control of a processor built into the electrical unit).

After the formation is removed, the resection site is examined in white light, then virtual chromoscopy (NBI), and then an examination with magnification. The examination results are recorded in the scientific protocol separately and are assessed as a whole. The criteria for visual removal of a lesion within healthy tissues are the absence of visible fragments of the lesion. The time until capillary bleeding completely stops is recorded.

If residual tissue of the lesion is detected, it is removed using the same technique. If the removal of residual tissue of the lesion was performed by another method, indicate which one ahnd why.

After Hot EMR , in half of the cases (according to the instructions of the randomized recording), "Australian" electroablation of the wound edges is performed with the tip of the polypectomy loop.

The removed lesion (all fragments) is extracted through the endoscope channel (for example, by aspiration) or by another method. The specimen not sent for morphological examination is considered lost.

Terminology (complications). Complications (adverse events) will be considered as occurring during the intervention (intraoperative), if they develop from the moment the colonoscope is inserted until it is removed. Otherwise, complications will be regarded as postoperative.

Perforation during the examination is diagnosed when the "target" symptom is detected - the presence of an additional ring-shaped structure at the bottom of the wound and/or during endoscopic visualization through defect of the organ wall.

Delayed perforation will be defined as the development of symptoms of peritoneal irritation and free gas in the abdominal cavity in the patient and/or the detection of a perforation hole in the area of removal of the formation during surgical revision.

Immediate bleeding is bleeding that has not stopped within 4 minutes (the normal hemostasis for capillary bleeding /from a finger/ according to Duke: onset after 2 minutes, end after 4 minutes) after removal of the formation and requiring one of the methods of endoscopic hemostasis (injection of adrenaline solution and/or coagulation (including ARS) and/or clipping.

Delayed bleeding is blood in the stool and unstable vital signs and/or a drop in hemoglobin ≥ 2 g / dl.

Postcoagulation syndrome is defined as the presence of abdominal pain and/or leukocytosis and/or fever (more than 37.2) and/or symptoms of peritoneal irritation in the case of:

1. The absence of these symptoms before the manipulation and other reasons for their appearance
2. The absence of free gas in the abdominal cavity and/or detection of a perforation in the area of removal of the formation during surgical revisions.

Methodology of morphological examination of preparations. After the preparation is extracted, it is fixed in a straightened state on thick adhesive paper or on a cork. In case of removal of the formation in fragments, the extracted fragments are also fixed in the above-mentioned manner. After fixation, the preparation is placed in a 10% formalin solution and delivered to the pathology department. After 24 hours of fixation, the preparation is removed from the formalin. Then the size of the formation is measured and parallel sections are made every 2-3 mm, which are placed in cassettes and undergo a standard procedure for preparing paraffin blocks, after which paraffin sections are made every 3-4 μm and a routine procedure for staining with hematoxylin and eosin. During the histological description of the preparation, it is planned to note the following parameters: number of fragments; size of the formation; its morphological type and differentiation; presence of a muscular plate of the mucosa, presence and thickness of the tissues of the submucosal layer, diameter of the largest vessel in the sample; presence of tissues of the formation along the horizontal and vertical borders formation.

R0 means the absence of formation cells along the border (vertical and horizontal) of the coagulation line (in Cold) or the removal line (in Hot).

Morphological classification of the formation will be carried out according to the WHO classification and the Vienna classification (see appendix).

When evaluating biopsies from the edges of the wound, the fact of the presence/absence of residual tissues of the formation (adenoma and/or adenocarcinoma and/or serrated formation) in the biopsy is indicated.

The morphologist is not informed about the method of removal (Cold or Hot) of the formation.

Registration of documentation and computer statistical processing of data. A separate medical card will be filled out for each patient in a closed database on the Internet.

Mandatory - endophotographs of the formation before its removal and the wound after the end of the intervention, allowing to evaluate the parameters included in the analysis.

Statistical processing of the obtained data will be carried out by the method of variation statistics with the calculation of the arithmetic mean, standard deviation, standard error of the mean and reliability criterion (p). Differences at a significance level of 95% at p<0.05 are considered reliable. In order to check the significance of the difference between the means in different groups by comparing the variances of these groups, it is planned to use the methods of ANOVA (from the English ANalysis Of VAriance). The Pearson correlation coefficient will be calculated to assess the presence or absence of a linear relationship between two variables and the tightness of this relationship. The calculations are planned to be made using the statistical section of the Microsoft Office Excel spreadsheet software package.

ELIGIBILITY:
Inclusion Criteria:

* A patient with one benign non-invasive epithelial formation of the colon of type Is and II, measuring 10-14 mm
* Age ≥ 18 years.
* Signed informed voluntary consent for colonoscopy and removal of formations using the methods under study.

Exclusion Criteria:

* Reasonable suspicion of severe dysplasia/cancer, including with submucosal invasion based on the results of preoperative assessment (NICE - 3; JNET - 2b and 3; Kudo - Vi and Vn).

  -. Colonic lesions less than 10 mm
* Recurrent lesion.
* Presence of widespread malignant tumour in any part of the colon.- Use of other methods of endoscopic removal of the lesion.
* IBD.
* Patient on haemodialysis
* Uncorrectable coagulopathy (INR> 1.5).
* Refusal to participate in the study.
* General contraindications to endoscopic examination.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-25 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Radicality of removal | 1 months after removal
  Based on the pathomorphological report, the radicality of the removal of the epithelial formation by the EMR and ESD methods will be assessed. (R0, R1, Rx)
Duration of the operation | at the time of the operation
  from the moment of submucosal injection until the complete removal of the formation, the duration of the operation will be recorded
Intraoperative complications | at the time of the operation
  During the operation, intraoperative complications that arise are recorded: perforation, bleeding
Postoperative complications | 1 months after removal
  Postoperative complications that arise from 1 day to 30 days after removal are assessed: postcoagulation syndrome, bleeding, perforation.
Relapse of education | 12 months after removal
  The postoperative scar is assessed for the presence of recurrent formation
Successful removal | at the time of the operation
  Analysis of the possibility of removal and the number of fragments

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny Gorbachev, Study Chair — Pirogov Russian National Research Medical University
Locations (1):
- Evgeny Gorbachev, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No